CLINICAL TRIAL: NCT01313481
Title: A Randomized Controlled Trial of the Effect of Otago Exercise Delivered as Home Exercise or Group Exercise in Fall-prone Older Persons
Brief Title: Effect of the Otago Programme Delivered as Home Exercise or Group Exercise
Acronym: FALLFOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other); Norwegian Fund for Postgraduate Training in Physiotherapy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6.2008.1352
Record Dates: First submitted 2010-03-22; First posted 2011-03-11 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Accidental Falls; Distorted Balance
Keywords: Older persons; Exercise; Balance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group exercise (Experimental): Otago exercise performed in groups
  Interventions: Behavioral: Group exercise
- Home exercise (Active Comparator): Otago exercise performed as home exercise
  Interventions: Behavioral: Home exercise

INTERVENTIONS:
Behavioral: Group exercise — Otago exercise performed in groups of 4-8 patients, 2 times a week over 12 weeks
  Arms: Group exercise
Behavioral: Home exercise — Otago exercise performed as home exercise 3 times a weeks over 12 weeks. Individually tailored physical balance and muscle strength exercise
  Arms: Home exercise

SUMMARY:
The study aims to assess the effect on functional balance of Otago exercise performed as home exercise versus group exercise. The investigators hypothesize that Otago exercise is more effective performed as group exercise than home exercise.

DETAILED DESCRIPTION:
The study sample is drawn from persons referred to a falls outpatient clinic. Group exercise and home exercise are delivered by trained physiotherapists. Home exercise follows the original Otago exercise protocol. Group exercise is performed twice a week. The length of the intervention period is 3 months. The main outcome measure is the Berg Balance Scale.

ELIGIBILITY:
Inclusion Criteria:

* referred to an outpatient falls clinic
* have fallen previous year or have gait or balance problems

Exclusion Criteria:

* Mini Mental Status Examination (MMSE) < 22
* Not able to walk 10 m without support from another person

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 125 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Functional Balance by use of the Berg Balance Scale | 3 months

SECONDARY OUTCOMES:
Fear of falling by the Fall Efficacy Scale International (FES-I), 7 item version | 3 and 6 months
Mobility by the Timed Get up-and-go | 3 and 6 months
Functional leg muscle strength by a Sit-to-stand test | 3 and 6 months
  Number of raise-up trials in 30 sec, picked from the Senior Fitness test
Health related quality of life by the Short Formular 36 (SF-36) | 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn L Helbostad, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Vestfold hospital, Tønsberg, Vestfold, Norway

REFERENCES:
- [Result] Kyrdalen IL, Moen K, Roysland AS, Helbostad JL. The Otago Exercise Program performed as group training versus home training in fall-prone older people: a randomized controlled Trial. Physiother Res Int. 2014 Jun;19(2):108-16. doi: 10.1002/pri.1571. Epub 2013 Dec 11. PMID 24339273